CLINICAL TRIAL: NCT03319914
Title: Observational Follow-up to ST-001 Calciphylaxis Pain Treatment With Intravenous Sodium Thiosulfate
Acronym: OF-CALISTA
Status: Terminated | Type: Observational
Why Stopped: Subjects did not receive Hope Pharmaceuticals' Sodium Thiosulfate Injection.
Sponsor: Hope Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: ST-003
Record Dates: First submitted 2017-10-20; First posted 2017-10-24 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-06

CONDITIONS: Calciphylaxis
Keywords: calciphylaxis, calcific uremic arteriolopathy,; calcium metabolism disorders; metabolic diseases; sodium thiosulfate
MeSH Terms: conditions — Calciphylaxis; Calcium Metabolism Disorders; Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ST-003 Observational: Calciphylaxis patients who participated in the ST-001 CALISTA

SUMMARY:
This is an 8-week observational follow-up study of patients who participated in the ST-001 CALISTA study (A Phase 3, Intravenous Sodium Thiosulfate for Acute Calciphylaxis Treatment: A Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial).

DETAILED DESCRIPTION:
This is an 8-week observational follow-up study of patients who participated in the ST-001 CALISTA study. In this ST-003 (OF-CALISTA) study, the occurrence of delayed adverse events, standard of care treatments for calciphylaxis (medications [including Sodium Thiosulfate Injection and pain medication], wound debridement, amputation, hyperbaric oxygen therapy, and surgical parathyroidectomy), and calciphylaxis-related complications (new or worsening skin lesions, ulceration, infection, sepsis and hospitalizations) will be recorded during an 8-week observation period following patient participation in the ST-001 CALISTA study (A Phase 3, Intravenous Sodium Thiosulfate for Acute Calciphylaxis Treatment: A Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial).

ELIGIBILITY:
Inclusion Criteria:

* Previously enrolled as a patient in ST-001 CALISTA study
* Willing to provide written informed consent
* Willing and able to adhere to all study-related procedures
* Willing to authorize release of medical records
* Willing to authorize collection of medical data from health care providers
* Provide email, home address and phone number where he/she can be reached

Exclusion Criteria:

• Patient did not participate in ST-001 CALISTA study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those calciphylaxis patients that previously participated in the ST-001 CALISTA study (A Phase 3, Intravenous Sodium Thiosulfate for Acute Calciphylaxis Treatment: A Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial).
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2018-11-09 (Actual); Study Completion 2018-11-09 (Actual)

PRIMARY OUTCOMES:
Observation of delayed adverse events, standard of care treatments for calciphylaxis following participation in ST-001 | 8 weeks
  Record the occurrence of delayed adverse events, standard of care treatments for calciphylaxis(medications [including Sodium Thiosulfate Injection and pain medication], wound debridement, amputation, hyperbaric oxygen therapy, and surgical parathyroidectomy), and calciphylaxis-related complications (new or worsening skin lesions, ulceration, infection, sepsis and hospitalizations) following participation in ST-001

CONTACTS AND LOCATIONS:
Overall Officials: Craig Sherman, MD, Study Director — Hope Pharmaceuticals
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Veterans Administration Medical Center, Albany, New York
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Undecided